CLINICAL TRIAL: NCT00002475
Title: A Trial of Active Intralymphatic Immunotherapy With Interferon-Treated Cells and Cyclophosphamide
Brief Title: Cyclophosphamide Plus Vaccine Therapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Vincent Medical Center - Los Angeles (Other)
Responsible Party: Charles L. Wiseman
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SVMC-ONC-222; CDR0000076913 (Registry Identifier: PDQ (Physician Data Query)); NCI-V91-0075
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Kidney Cancer; Lung Cancer; Malignant Mesothelioma; Pancreatic Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IIIC breast cancer; stage IV non-small cell lung cancer; pulmonary carcinoid tumor; recurrent malignant mesothelioma; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Mesothelioma, Malignant; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Small Cell Lung Carcinoma | interventions — FANG vaccine; Interferon-alpha; Interferon-gamma; sargramostim; Cyclophosphamide

INTERVENTIONS:
Biological: allogeneic tumor cell vaccine
Biological: autologous tumor cell vaccine
Biological: recombinant interferon alfa
Biological: recombinant interferon gamma
Biological: sargramostim
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Vaccines made from a patient's tumor tissue may make the body build an immune response to kill tumor cells. Chemotherapy combined with vaccine therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining cyclophosphamide with tumor cell vaccine in treating patients who have metastatic cancer or cancer at high risk of recurrence.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and clinical effects of autologous or allogeneic active-specific intralymphatic immunotherapy with a vaccine containing interferon alfa or interferon gamma-treated tumor cells followed by sargramostim (GM-CSF) in patients with advanced cancer.

OUTLINE: This is a pilot study. Patients are stratified by tumor type.

Tumor tissue is removed from the patient and incubated with interferon alfa or interferon gamma for 72-96 hours. (If autologous tumor cells are not available, an allogeneic vaccine is prepared.) Harvested activated cells are irradiated immediately prior to use.

Patients receive cyclophosphamide IV. 48-72 hours after cyclophosphamide administration, patients receive tumor cell vaccine intradermally. Patients also receive sargramostim (GM-CSF) subcutaneously prior to vaccine administration and once daily for the next 8 days. Treatment repeats every 2 weeks for 3 courses in the absence of unacceptable toxicity. Patients with responding or stable disease after completion of course 3 may receive additional courses.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer not amenable to cure or long-term control by surgery, radiotherapy, chemotherapy, or hormonal manipulations, including the following tumor types:

  * Colon cancer
  * Lung cancer
  * Renal cancer
  * Breast cancer
  * Pancreatic cancer
* Metastatic disease or subclinical disease at high risk of recurrence
* No brain metastases unresponsive to irradiation or surgery
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No prior or concurrent significant cardiovascular disease

Pulmonary:

* No prior or concurrent pulmonary disease

Other:

* No prior or concurrent autoimmune disease
* No other prior or concurrent major medical illness
* HIV negative
* No clinical evidence of AIDS
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hormonal therapy
* No concurrent chronic steroid therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1991-04; Primary Completion 2007-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical response (patients with evaluable disease)
Duration of response (patients with evaluable disease)
Survival (patients with evaluable disease)
Time to recurrence (patients without evaluable disease)
Survival (patients without evaluable disease)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Wiseman, MD, FACP, Study Chair
Locations (1):
- St. Vincent Medical Center - Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Wiseman C, Presant C, Rao R, Smith J. Clinical responses to intralymphatic whole-cell melanoma vaccine augmented by in vitro incubation with alpha-interferon. Ann N Y Acad Sci. 1993 Aug 12;690:388-91. doi: 10.1111/j.1749-6632.1993.tb44040.x. No abstract available. PMID 8368765